CLINICAL TRIAL: NCT01332526
Title: The Oral Fructose Load Test and Inflammation, Lipid Metabolism, Blood Pressure and Organ Damage in Patients With Obesity, Chronic Kidney Disease With Comparison With Healthy Controls.
Brief Title: FFT, Inflammation, Lipid Metabolism, Blood Pressure and Organ Damage in Patients With Obesity, Chronic Kidney Disease (CKD).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Richard Johnson M.D., Chief, Division of Renal Diseases and Hypertension
Other Study IDs: FFT Bydgoszcz
Record Dates: First submitted 2011-03-31; First posted 2011-04-11 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-03

CONDITIONS: Obesity; Chronic Kidney Disease; Metabolic Syndrome
Keywords: FFT; inflammation; lipid metabolism; hyperuricemia; Agents Affecting Uric Acid Metabolism
MeSH Terms: conditions — Obesity; Renal Insufficiency, Chronic; Metabolic Syndrome; Inflammation; Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (7):
- Patients with BMI> 30 and metabolic syndrome ( ATP III).: Patients with BMI> 30 and metabolic syndrome ( ATP III).
- Patient with BMI> 30 without metabolic syndrome.: Patient with BMI> 30 without metabolic syndrome.
- Normal healthy control: healthy persons( without renal disease, cardiovascular diseases, diabetes mellitus, BMI < 25;normotensives ).
- Patients with CKD stage III and uric acid < 7 mg/dl: Patients with CKD stage III (GFR 30-59 ml/min/1,73 m2) and uric acid < 7 mg/dl.
  * without diabetes mellitus proteinuria < 3,5 g/24 h without immunosuppressives agents, ACEi, ARB, allopurinol treatment well controlled hypertension ( < 140/90 mmHg)
- Patients with CKD stage III and uric acid > 7 mg/dl: Patients with CKD stage III(GFR 30-59 ml/min/1,73 m2) and uric acid > 7 mg/dl
  * without diabetes mellitus proteinuria < 3,5 g/24 h without immunosuppressive agents, ACEi, ARB, allopurinol treatment well controlled hypertension ( < 140/90 mmHg)
- Patient with asymptomatic hyperuricemia: Patient with asymptomatic hyperuricemia, uric acid > 7 mg/dl with normal renal function
- Hemodialysis patients: Patient with asymptomatic hyperuricemia, uric acid > 7 mg/dl with normal renal function Hemodialysis patients.
  * CKD: nondiabetic nephropathy
  * duration hemodialysis 3-48 months
  * Hb-11-13 g/dl
  * well controlled hypertension ( < 140/90 mmHg)
  * without ACEi, ARB, allopurinol treatment
  * residual diuresis will be estimated for last 48 hours-between mid and next dialysis

SUMMARY:
Fructose intake from added sugars has increased dramatically over the last century and has recently been implicated as potential contributor to metabolic syndrome, obesity, hypertension, inflammation and kidney disease. Fructose differs from the other sugars because, uric acid is generated during its metabolism. Serum uric acid levels have been found to correlate with the intake of fructose and added sugars. In turn, an elevated serum uric acid has also been shown to be associated with increased risk for cardiovascular and metabolic diseases. On the other hand complexity of fructose metabolism in each individuals results of the various magnitude of hyperuricemia induced by fructose intake. The magnitude of uric acid production in each patient may reflect individual predisposition to endogenous urate production in a face of relatively normal fasting uric acid concentration. Therefore the oral fructose tolerance test might reveal an occult purine disturbances which plays casual role in either metabolic disturbances or organ damage.

The aim of this study is to see whether is a relationship between fructose induced hyperuricemia and metabolic disturbances , inflammatory state and organ damage in obese and various stages CKD patients.

DETAILED DESCRIPTION:
The study will be performed in two experimental groups. Proposed study groups Study I Patients with BMI> 30 and metabolic syndrome. Patient with BMI> 30 without metabolic syndrome. Normal healthy controls. Study II Patients with CKD stage III and uric acid < 7 mg/dl Patients with CKD stage III and uric acid > 7 mg/dl Patient with asymptomatic hyperuricemia and eGFR > 90 ml/min/1.73 m2, , uric acid > 7 mg/dl Hemodialysis patients

Characteristics of the particular patients group- including criteria:

10- 15 participants in each subset of each group age 18-65 y. Gender: females and males in equal proportion. Group I Patients with BMI> 30 and metabolic syndrome ( ATP III). Patient with BMI> 30 without metabolic syndrome. Normal healthy control- healthy persons( without renal disease, cardiovascular diseases, diabetes mellitus, BMI < 25;normotensives ).

Group II Patients with CKD stage III (GFR 30-59 ml/min/1,73 m2) and uric acid < 7 mg/dl.

* without diabetes mellitus proteinuria < 3,5 g/24 h without immunosuppressive agents, ACEi, ARB, allopurinol treatment well controlled hypertension ( < 140/90 mmHg) Patients with CKD stage III(GFR 30-59 ml/min/1,73 m2) and uric acid > 7 mg/dl
* without diabetes mellitus proteinuria < 3,5 g/24 h without immunosuppressive agents, ACEi, ARB, allopurinol treatment well controlled hypertension ( < 140/90 mmHg)

Patient with asymptomatic hyperuricemia, uric acid > 7 mg/dl with normal renal function Hemodialysis patients.

* CKD: nondiabetic nephropathy
* duration hemodialysis 3-48 months
* Hb-11-13 g/dl
* well controlled hypertension ( < 140/90 mmHg)
* without ACEi, ARB, allopurinol treatment
* residual diuresis will be estimated for last 48 hours-between mid and next dialysis Method of investigation All patients and controls ( but hemodialysis) will present after overnight fast. Baseline tests include 24 hr urine collection for: sodium, calcium, phosphorus, creatinine, uric acid, NAG, albumin will be carry out and the same morning fasting sample of blood for: creatinine, cystatin C , uric acid, sodium, glucose, insulin, triglycerides, HDL and LDL cholesterol, calcium, phosphorus, hsCRP. BP will be determined as the mean of three readings taken 5 min apart while sitting. Next in all patients and controls fructose tolerance test will be performed. The test consists of giving 1 gram/kg b.w. of fructose p.o. with blood collection at 0,30,60 and 120 min afterward for serum uric acid determination and uric acid area under the curve will be calculated. The calculated area under curve is the measure of occult uric acid disturbance when compared to controls.

Day before the urine collection the ABPM , BMI, IM (intima media ratio) , renal duplex ultrasound (RI) will be done

Measure BMI, waist circumference

ELIGIBILITY:
Inclusion Criteria:

- Group I Patients with BMI> 30 and metabolic syndrome ( ATP III). Patient with BMI> 30 without metabolic syndrome. Normal healthy control- healthy persons( without renal disease, cardiovascular diseases, diabetes mellitus, BMI < 25;normotensives ).

Group II Patients with CKD stage III (GFR 30-59 ml/min/1,73 m2) and uric acid < 7 mg/dl.

* without diabetes mellitus proteinuria < 3,5 g/24 h without immunosuppressives agents, ACEi, ARB, allopurinol treatment well controlled hypertension ( < 140/90 mmHg) Patients with CKD stage III(GFR 30-59 ml/min/1,73 m2) and uric acid > 7 mg/dl
* without diabetes mellitus proteinuria < 3,5 g/24 h without immunosuppressive agents, ACEi, ARB, allopurinol treatment well controlled hypertension ( < 140/90 mmHg)

Patient with asymptomatic hyperuricemia, uric acid > 7 mg/dl with normal renal function Hemodialysis patients.

* CKD: nondiabetic nephropathy
* duration hemodialysis 3-48 months
* Hb-11-13 g/dl
* well controlled hypertension ( < 140/90 mmHg)
* without ACEi, ARB, allopurinol treatment
* residual diuresis will be estimated for last 48 hours-between mid and next dialysis

Exclusion Criteria:

* immunosuppressive agents, ACEi, ARB, allopurinol treatment
* diabetes mellitus
* not well controlled hypertension ( > 140/90 mmHg)
* proteinuria > 3,5 g/24 h

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study I Patients with BMI> 30 and metabolic syndrome. Patient with BMI> 30 without metabolic syndrome. Normal healthy controls. Study II Patients with CKD stage III and uric acid < 7 mg/dl Patients with CKD stage III and uric acid > 7 mg/dl Patient with asymptomatic hiperuricemia and eGFR > 90 ml/min/1.73 m2, , uric acid > 7 mg/dl Hemodialysis patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-05

CONTACTS AND LOCATIONS:
Overall Officials: Jacek JM Manitius, Study Chair — Department of Nephrology, Hypertension and Internal Diseases Nicolaus Copernicus University in Torun Poland Collegium Medicum in Bydgoszcz

REFERENCES:
- [Derived] Donderski R, Miskowiec-Wisniewska I, Kretowicz M, Grajewska M, Manitius J, Kaminska A, Junik R, Siodmiak J, Stefanska A, Odrowaz-Sypniewska G, Pluta A, Lanaspa M, Johnson RJ. The fructose tolerance test in patients with chronic kidney disease and metabolic syndrome in comparison to healthy controls. BMC Nephrol. 2015 May 3;16:68. doi: 10.1186/s12882-015-0048-y. PMID 25935771